CLINICAL TRIAL: NCT06009042
Title: Efficacy of Intravenous Immunoglobulin in Patients With Hemorrhagic Fever With Renal Syndrome: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Efficacy of Intravenous Immunoglobulin in Patients With Hemorrhagic Fever With Renal Syndrome: a Prospective Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director, Department of Infectation, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMISE
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: HFRS (Hemorrhagic Fever With Renal Syndrome)
Keywords: efficacy; IVIG（intravenous immunoglobulin）
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIG 20g/d (Experimental): Participants will receive IVIG (intravenous immunoglobulin) 20g/d for 6 days. They also receive conventional liquid therapy and symptomatic supportive treatment.
  Interventions: Drug: IVIG 20g/d
- IVIG 10g/d (Active Comparator): Participants will receive IVIG (intravenous immunoglobulin) 10g/d for 6 days. They also receive conventional liquid therapy and symptomatic supportive treatment.
  Interventions: Drug: IVIG 10g/d

INTERVENTIONS:
Drug: IVIG 20g/d — The dose of IVIG(intravenous immunoglobulin) is 20g/d. Participants also receive conventional liquid therapy and symptomatic and supportive treatment.
  Arms: IVIG 20g/d
Drug: IVIG 10g/d — The dose of IVIG(intravenous immunoglobulin) is 10g/d. Participants also receive conventional liquid therapy and symptomatic and supportive treatment.
  Arms: IVIG 10g/d

SUMMARY:
The goal of this randomized study to test the efficacy of different doses of IVIG (intravenous immunoglobulin) in the treatment of severe HFRS（hemorrhagic fever with renal syndrome）, and provide new clinical ideas for the treatment and prognosis of HFRS patients in the future.

This study will include all hospitalized patients with confirmed severe or critically ill HFRS from October 2021 to October 2023 from 9 centers.

Participants will receive IVIG 10g/d or IVIG 20g/d. All the participants will be given conventional liquid therapy and symptomatic and supportive treatment.

Participants will be collected demographic, epidemiological history, hospitalization information, clinical data, laboratory data, imaging results, treatment regimens, and outcomes data.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized controlled study which aims at evaluating the efficacy of different doses of IVIG (intravenous immunoglobulin) in the treatment of patients with severe HFRS(hemorrhagic fever with renal syndrome), and providing reference for the future application of IVIG in severe hemorrhagic fever with renal syndrome. This study will include approximately 100 patients with severe hemorrhagic fever with renal syndrome who are randomly assigned to either the IVIG 10g/d group or the IVIG 20g/d group in a 1:1 ratio. The participants in each group will receive treatments for 6 days. Both groups are given routine liquid therapy and symptomatic supportive treatment. The main endpoints include transformation rate, post-period rate, mortality rate, and duration of the disease. Secondary endpoints include the incidence of complications and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

The patients must meet all of the following criteria:

* Age ≥ 18 years, regardless of gender;
* Within 5 days of onset, hospitalized patients diagnosed with epidemic hemorrhagic fever (hemorrhagic fever with renal syndrome) must have at least one of the following laboratory test results:

  1. Positive for serum specific IgM(immunoglobulin M) antibodies;
  2. Or detect hantavirus RNA(ribonucleic acid) from patient specimens;
  3. Or the serum specific IgG(immunoglobulin G) antibody titer in the recovery phase is more than four times higher than that in the acute phase;
  4. Or hantavirus can be isolated from patient specimens.
* Meet any of the following criteria:

  1. Severe illness: meet any of the following criteria: (i) Platelet count 20-50×10^9/L; (ii) White blood cell count 15-30×10^9/L. 2. Critical illness: meet any of the following criteria: (i) Platelet count<20×10^9/L; (ii) White blood cell count>30×10^9/L.
* Volunteer to join this study and be able to sign or have a written informed consent form signed by a legal representative.

Exclusion Criteria:

Exclude patients who meet any of the following criteria:

* Patients with primary chronic kidney disease;
* Patients with severe diabetes, hypertension, heart, lung, gastrointestinal tract, liver, autoimmune disease or nervous system disease;
* Have a history of malignant tumors (including solid malignant tumors and hematological malignancies etc.);
* Recent use of potentially nephrotoxic drugs;
* Pregnant or potentially pregnant patients;
* Patients with a history of hypersensitivity to IVIG (intravenous immunoglobulin) ;
* Selective IgA(immunoglobulin A) deficiency patients with IgA antibodies;
* Known or suspected immunodeficiency (human immunodeficiency virus infection, primary immunodeficiency), use of immunosuppressive drugs (glucocorticoids);
* Alcoholics, drug abuse, and psychiatric patients
* Other conditions which researchers deem not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Transformation rate | up to 34th day after treatment
  The transformation rate is defined as the rate of transformation [critical to severe, moderate or mild, severe to moderate or mild], or the rate of transition [severe to critical].
Post-period rate | up to 34th day after treatment
  Post-period rate is defined as post-hypotension shock phase or oliguric phase, or post-hypotension shock phase and oliguric phase
Mortality rate | up to 34th day after treatment
The duration of the disease | up to 34th day after treatment
  The duration of the disease is defined as the duration from symptom onset to recovery and discharge.

SECONDARY OUTCOMES:
The incidence of complications | up to 34th day after treatment
  The incidence of complications is defined as the incidence of shock, renal failure, disseminated intravascular coagulation.
length of hospital stay | up to 34th day after treatment
  The length of hospital stay is defined as the number of days from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Professor, Principal Investigator — Tongji Hospital
Locations (9):
- China (9):
  - No.1 Peoples Hospital of Guangshui, Guangshui, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - People's Hospital of Luotian County, Huanggang, Hubei
  - People's Hospital of Macheng City, Affiliated Hospital of Hubei University of Science and Technology, Macheng, Hubei
  - Qianjiang Central Hospital, Qianjiang, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - The Third Peoples Hospital of Yichang, Yichang, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu